CLINICAL TRIAL: NCT01099969
Title: Endotrol-tracheal Tube Assisted Endotracheal Intubation During Video Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Davide Cattano, Associate Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-09-0456
Record Dates: First submitted 2010-04-01; First posted 2010-04-08 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Endotracheal Intubation
Keywords: Endotrol Endotracheal tube; Regular endotracheal tube; gliderite stylet; McGrath videolaryngoscope; Glidescope

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glidescope with non-styletted Endotrol ETT (Experimental): The patients in this arm will be intubated using a Glidescope videolaryngoscope with non-styletted Endotrol endotracheal tube (ETT).
  Interventions: Device: Glidescope videolaryngoscope; Device: Non-styletted Endotrol endotracheal tube (ETT)
- Glidescope with styletted regular ETT (Active Comparator): The patientsin this arm will be intubated using the glidescope videolaryngoscope and regular endotracheal tube (ETT) with gliderite stylet.
  Interventions: Device: Glidescope videolaryngoscope; Device: Regular endotracheal tube (ETT) with Gliderite stylet
- McGrath with non-styletted Endotrol ETT (Experimental): The patients in this arm will be intubated using McGrath videolaryngoscope and non-styletted Endotrol endotracheal tube (ETT).
  Interventions: Device: McGrath videolaryngoscope; Device: Non-styletted Endotrol endotracheal tube (ETT)
- McGrath with with styletted regular ETT (Active Comparator): The patients receiving this arm will be intubation using McGrath videolaryngoscope and regular endotracheal tube (ETT) with Gliderite stylet.
  Interventions: Device: McGrath videolaryngoscope; Device: Regular endotracheal tube (ETT) with Gliderite stylet

INTERVENTIONS:
Device: Glidescope videolaryngoscope
  Arms: Glidescope with non-styletted Endotrol ETT; Glidescope with styletted regular ETT
Device: McGrath videolaryngoscope
  Arms: McGrath with non-styletted Endotrol ETT; McGrath with with styletted regular ETT
Device: Non-styletted Endotrol endotracheal tube (ETT)
  Arms: Glidescope with non-styletted Endotrol ETT; McGrath with non-styletted Endotrol ETT
Device: Regular endotracheal tube (ETT) with Gliderite stylet
  Arms: Glidescope with styletted regular ETT; McGrath with with styletted regular ETT

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Endotrol Tube compared to the conventional endotracheal tube in conjunction with the GlideRite stylet (Verathon Medical Inc, USA) during videolaryngoscopy assisted endotracheal intubation using a McGrath (Aircraft Medical Ltd., and distributed in the US by LMA North America, Inc.) video laryngoscope or a GlideScope (Verathon Medical Inc, USA). The investigators hypothesize that using the Endotrol tracheal tube, (Covidien, Colorado, USA) is safer and more efficacious than using the conventional endotracheal tube during McGrath video laryngoscope and/or GlideScope aided endotracheal intubation.

DETAILED DESCRIPTION:
It is estimated that endotracheal intubation is performed on some 8 million patients per year in the United States. Of these endotracheal intubations, approximately 80% are performed by direct laryngoscopy with transoral placement of the endotracheal tube (ET) into the trachea. There is fairly uniform reporting of the incidence of failed intubation in the literature; it occurs in approximately 0.05% or 1:2230 of surgical patients and in approximately 0.13% to 0.35%, or 1:750 to 1:280, of the obstetric patients.1,2 The incidence of unsuspected difficult intubation is estimated to be higher at 3%. One factor that contributes to difficult intubation is poor visualization of the airway. Video laryngoscopes are a relatively new edition to the armamentarium of airway devices available to the airway manager. Although these instruments are more expensive than traditional direct laryngoscopes, they offer several advantages that may justify their expense. Although some clinicians may espouse the routine use of video laryngoscopy, most providers reserve it for anticipated difficult situations or as "plan B" after failed intubation by direct laryngoscopy (DL). There are several advantages of a video intubation technique as compared to direct laryngoscopy. The video laryngoscopes have been shown to provide superior views to traditional laryngoscopy as well as in difficult intubations.3-5 Video intubation techniques, by allowing tracheal intubation monitoring, have been shown to improve the safety of the procedure and increase intubation success. The GlideScope consists of a digital camera, called a video baton, which fits into a plastic laryngoscope blade and a light source on the side to provide a video image of airway structures on a screen, which can be conveniently located directly in front of the anesthesiologist. The GlideRite rigid stylet conforms to the GlideScope blade angulation, which,eliminates the need to manually shape the stylet to fit down the airway and improves maneuverability in endotracheal tube placement.

It should be noted that several reports have been published describing trauma to the upper airway (anterior tonsillar pillar, soft palate) during intubation with video laryngoscopes. Recently, several reports using endoflex tube (which is similar to the endotrol tube) showed that there is considerable usefulness in normal direct laryngoscopy and video laryngoscopy (using glidescope) as well. The purpose of this study is to compare the safety and efficacy of Endotrol Tube (Covidien, Colorado, USA) compared to the conventional endotracheal tube in conjunction with the GlideRite stylet during videolaryngoscopy assisted endotracheal intubation.

INSTRUMENTS:

McGrath Video Laryngoscope (MVL) - A video-based system for tracheal intubation that utilizes a video camera embedded into a "camera stick". The resulting video image is displayed on a small color Liquid Crystal Display (LCD) attached to the top of the handle of the device, which can be adjusted to obtain the best view. The unit is powered with a single easily-replaced AA battery and features a single electronic control: an on/off switch located on the top of the unit. The device is available with an adjustable curved MAC blade (sizes 3 to 5). Also,the device features a sterile disposable transparent blade sheath preventing cross infection.

GlideScope Video Laryngoscope (GVL)- The GlideScope was commercially introduced in 2001. The 1- piece handle and blade is made of medical- grade plastic. It has a vertical profile of 14.5 mm, a midblade bend of 50-60 degrees, and a video camera with a light-emitting diode housed toward the distal end of the blade. The image captured by the camera is transferred by the attached cable to a color liquid crystal display (LCD). A heating element covers the camera lens and ensures effective antifogging after the device has been turned on for 15- 30 seconds. The blades can be sterilized and reused, and are available in 3 sizes: large (adult), midsize (pediatric), and small (neonatal). As the image is transferred to the LCD display, anesthesiologists are able to view key anatomical landmarks at the earliest possible time, facilitating navigation. Also, in cases requiring external laryngeal manipulation, the assistant can see the effect of the maneuver on the monitor simultaneously with the anesthesiologist for quicker, more efficient intubation. Endotrol Tracheal Tube (ETT) (Covidien, Colorado, USA) - A sterile, single lumen, disposable ET with a built- in flexing mechanism with a standard 15 mm connector. The tube provides directional tip control via an operator- activated ring loop and incorporates a self- sealing valve with attached pilot balloon. The ETT is specifically designed for use in cases where difficult intubation can be aided with directional tip control. Due to the Hi-Lo cuff design, the ETT is acceptable for oral/nasal intubation of the trachea for anesthesia and in cases where the intubation duration is expected to be more than 24 hours or unpredictable. The special way to hold the ETT is to place the thumb of the right hand against the end of the 15 mm connector and the index finger in the ring loop. Pulling on the ring loop causes the tip to turn anteriorly towards the tracheal opening.

METHODOLOGY:

A. General Study Design- The study will include a total of 60 patients. Patients will be randomized into 2 groups and 2 subgroups in each group, through a computer generated randomization schedule.

Patients in group A (N= 30) will be intubated using MVL and patients in group B (N= 30) will be intubated using GVL. Patients in each group will be divided into 2 subgroups.

Group A (N= 30) - Subgroup A1 (N=15) - Patients will be intubated using Endotrol Tracheal Tube without stylet (Covidien, Colorado, USA). Subgroup A2 (N= 15) - Patients will be intubated using styletted endotracheal tube the Gliderite (Teleflex Medical, Hudson RCI/ Sheridan/ HBT). Group B (N= 30) - Subgroup B1 (N=15) - Patients will be intubated using Endotrol Tracheal Tube without stylet (Covidien, Colorado, USA).

. Subgroup B2 (N= 15) - Patients will be intubated using styletted endotracheal tube the Gliderite (Teleflex Medical, Hudson RCI/ Sheridan/ HBT). In the operating room, standard monitoring devices will be applied including a pulse oximeter, 3 lead (at least), ECG and blood pressure cuff; the latter could be invasive or non-invasive depending on the nature of the surgery. Baseline measures of BP, pulse, oxygen saturation, and CO2, will be made. The time will be noted before any sedation or anesthesia is administered. Vital signs will be recorded every minute from the time that induction of anesthesia is begun until five minutes after the patient has been intubated, and then at five-minute intervals thereafter for fifteen minutes. General anesthesia will be induced by bolus administration of propofol (2mg/kg) and fentanyl (1mcg/kg), and maintained with an inhalational agent. Rocuronium (0.6 mg/kg) will be administered to provide muscle relaxation and a mixture of sevoflurane or isoflurane and nitrous oxide will be utilized for maintenance of anesthesia once the ability to mask ventilate is confirmed. The lungs will be mechanically ventilated with a semi-closed circle system to maintain an end-tidal CO2 near 35 mmHg. Patients' lungs will be ventilated via anesthesia mask 100% oxygen until the patient is completely relaxed. All investigators will be trained based on manufacturer recommendations and each resident will perform at least 3 intubations with McGrath laryngoscope and 3 intubations with Cobalt GlideScope (total of 6 intubations) prior to enlisting any patients for the study. The CA-2 and CA-3 residents will be performing the intubations. The external neck pressure may be applied by an assistant in an attempt to improve exposure of the larynx. The ease of intubation will be recorded in terms of the number of attempts (measured as either the reinsertion of the blade or endotracheal tube) and the intubation time (time the laryngoscope blade enters the mouth until 1st capnograph breath) will be recorded. If more than 2 attempts were needed, a third attempt can be made with the device used in the other group. If still unsuccessful, the direct laryngoscopy/ flexible fibreoptic laryngoscopy will be performed to intubate the trachea and the case will be deemed a failure. The subjective level of difficulty (from 0 = Extremely Easy to 5 = Extremely Difficult) in the performance of intubation will also be recorded. An alternative technique will be used in case the intubation fails. 1. Use of the Glideride stylet if using an Endotrol tracheal tube, if the Endotrol tracheal tube is not able to get towards the cords. 2. Use of a regular stylet instead of the Glideride especially with McGrath if Glideride not able to help with intubation 3. Use of macintosh or miller appropriate blade with styletted or Endotrol tube if intubation with videolaryngoscope is difficult 4. Use of LMA or similar device in case intubation is difficult with any of the previous devices and application of a difficult airway protocol. B. Measurements- We will record morphometric characteristics of all patients. The quality of the airway will be evaluated using the Mallampati and Wilson scoring system, thyromental scoring system of Patil, interincisor gap distance, neck mobility and sternomental distance.

Additionally, the anesthesiologist will provide a personal, subjective opinion of a possible difficult intubation. Intubation: We will measure the time and number of attempts required for successful endotracheal intubation in each group. An attempt is defined as an attempt at placement of an ET through the glottic opening and into the trachea. Removal/reinsertion of the laryngoscope or the switching of the laryngoscopist will constitute as a new attempt. The subjective level of difficulty (0-5) in the performance of intubation will also be recorded. Once an optimal positional has been confirmed, position of the ET will not be further altered. Degree of irritation: Following intubation in either group, the appearance of oropharynx, pharynx, epiglottis, and arytenoids will be checked. The presence of abrasions, bleeding, redness, perforation or other signs of tissue or dental injury will be recorded.

SUBJECTS:

The subjects will be adult surgical candidates age 18-80, ASA I- III, presenting for elective surgery who require general anesthesia. Patients will be chosen if it is determined that endotracheal intubation is required. Patients will be excluded if they are considered so difficult (i.e. Mallampatti IV, < 2 FB or 4 cm mouth opening), that an awake fibreoptic intubation should be performed. ASA IV and V patients will also be excluded.

RECRUITMENT METHODS/ INFORMED CONSENT:

Physician investigators will interview all potential subjects to determine if subjects are suitable for the study. Both English and Spanish speaking subjects will be enrolled for the study. Written consent will be obtained by an anesthesiology resident or research assistant.

PROCEDURES TO MAINTAIN CONFIDENTIALITY:

All information recorded on the anesthetic records will be kept strictly confidential and all data will be kept in a data logbook locked in the office of the principal investigator. We will record patients only by study code number.

DATA ANALYSIS:

Data will be compared using two- tailed paired t- tests, repeated measures of ANOVA, or Fisher Exact test, as appropriate. Results will be presented as means ± SD. P < 0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old
* ASA: I-III
* Mallampati: I-III
* Mouthopening: 2 FB or < 4 cm

Exclusion Criteria:

* Age < 18 years or > 80 years
* ASA: IV
* Mallampati: IV
* Mouthopening < 2 FB 4cm
* No risk for aspiration
* No respiratory infection in past 10 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Cattano, M.D.,PhD, Principal Investigator — The University of Texas Medical School at Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GlideScope With Non-styletted Endotrol ETT: The patients in this arm will be intubated using a GlideScope videolaryngoscope with non-styletted Endotrol endotracheal tube (ETT).
  GlideScope videolaryngoscope
  Non-styletted Endotrol endotracheal tube (ETT)
- GlideScope With Styletted Regular ETT: The patients in this arm will be intubated using the GlideScope videolaryngoscope with regular endotracheal tube (ETT) with GlideRite stylet.
  GlideScope videolaryngoscope
  Regular endotracheal tube (ETT) with GlideRite stylet
- McGrath With Non-styletted Endotrol ETT: The patients in this arm will be intubated using McGrath videolaryngoscope and non-styletted Endotrol endotracheal tube (ETT).
  McGrath videolaryngoscope
  Non-styletted Endotrol endotracheal tube (ETT)
- McGrath With With Styletted Regular ETT: The patients receiving this arm will be intubation using McGrath videolaryngoscope and regular endotracheal tube (ETT) with GlideRite stylet.
  McGrath videolaryngoscope
  Regular endotracheal tube (ETT) with GlideRite stylet
Period: Overall Study
Arm/Group | GlideScope With Non-styletted Endotrol ETT | GlideScope With Styletted Regular ETT | McGrath With Non-styletted Endotrol ETT | McGrath With With Styletted Regular ETT
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GlideScope With Non-styletted Endotrol ETT | GlideScope With Styletted Regular ETT | McGrath With Non-styletted Endotrol ETT | McGrath With With Styletted Regular ETT | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (13.1) | 41.2 (14.4) | 50.4 (14.1) | 50.7 (15.7) | 49.5 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 7 | 7 | 32
  Male | 8 | 4 | 8 | 8 | 28
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Intubation Time
Description: Intubation time is the time from insertion of the laryngoscope to detection of CO2 on the capnogram.
Time Frame: time from insertion of the laryngoscope to detection of CO2 on the capnogram
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | GlideScope With Non-styletted Endotrol ETT | GlideScope With Styletted Regular ETT | McGrath With Non-styletted Endotrol ETT | McGrath With With Styletted Regular ETT
Number analyzed (Participants) | 15 | 15 | 15 | 15
seconds | 60.2 (34.8) | 48.8 (30.8) | 58.6 (29.9) | 40.7 (24.4)

2. Primary Outcome: Number of Intubation Attempts
Time Frame: at the time of placement of the endotracheal tube
Measure: Count of Participants; unit: Participants
Arm/Group | GlideScope With Non-styletted Endotrol ETT | GlideScope With Styletted Regular ETT | McGrath With Non-styletted Endotrol ETT | McGrath With With Styletted Regular ETT
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  1 attempt | 13 | 14 | 14 | 13
  2 attempts | 1 | 0 | 0 | 1
  3 attempts | 1 | 1 | 1 | 1

3. Primary Outcome: Number of Difficult Intubations
Description: Ease of intubation was subjectively assessed by the operator on a scale from 1 to 5 (1 = extremely easy, 2 = easy, 3 = neutral, 4 = difficult, 5 = extremely difficult). A score of 4 or 5 was characterized as "difficult."
Time Frame: at the time of placement of the endotracheal tube
Measure: Number; unit: intubations
Arm/Group | GlideScope With Non-styletted Endotrol ETT | GlideScope With Styletted Regular ETT | McGrath With Non-styletted Endotrol ETT | McGrath With With Styletted Regular ETT
Number analyzed (Participants) | 15 | 15 | 15 | 15
intubations | 1 | 0 | 2 | 0

4. Secondary Outcome: Cormack and Lehane Grade of Laryngeal View
Description: The Comarck Lehane classification is as follows: 1)Full view of glottis; 2a) Partial view of glottis; 2b) Only posterior extremity of glottis seen or only arytenoid cartilages; 3) only epiglottis is seen, none of glottis seen; 4) neither glottis nor epiglottis seen.
Time Frame: at the time of intubation
Measure: Count of Participants; unit: Participants
Arm/Group | GlideScope With Non-styletted Endotrol ETT | GlideScope With Styletted Regular ETT | McGrath With Non-styletted Endotrol ETT | McGrath With With Styletted Regular ETT
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  1 | 12 | 11 | 13 | 13
  2a | 2 | 4 | 1 | 1
  2b | 1 | 0 | 1 | 1
  3 | 0 | 0 | 0 | 0
  4 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: On the day of surgery
Arm/Group | GlideScope With Non-styletted Endotrol ETT | GlideScope With Styletted Regular ETT | McGrath With Non-styletted Endotrol ETT | McGrath With With Styletted Regular ETT
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
small sample size; study not controlled for the residents' personal experience, and some performed more intubations compared to others; ease of intubation was assessed subjectively by the operator who was unblinded to the modality used.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes